CLINICAL TRIAL: NCT01214187
Title: Phase II Study of Inhaled CO for the Treatment of Idiopathic Pulmonary Fibrosis
Brief Title: Study of Inhaled Carbon Monoxide to Treat Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of California, San Francisco (Other); University of Chicago (Other); University of Illinois at Chicago (Other); University of Michigan (Other); Columbia University (Other); Tulane University (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Ivan O. Rosas, Overall Principle Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1U01HL105371 (NIH); 1U01HL105371 (NIH)
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis; IPF; pulmonary fibrosis; carbon monoxide
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carbon monoxide inhalation (Experimental): The primary intervention will be inhaled CO at 100-200 ppm administered two times weekly for two hours per dose to complete 12 weeks of treatment.
  Interventions: Drug: inhaled carbon monoxide
- Oxygen 21% (Placebo Comparator)
  Interventions: Other: Oxygen

INTERVENTIONS:
Drug: inhaled carbon monoxide — The intervention will be inhaled CO at 100-200 ppm administered two times weekly for two hours per dose to complete 12 weeks of treatment.
  Other Names: CO
  Arms: carbon monoxide inhalation
Other: Oxygen — Room air oxygen concentrations will be administered as placebo
  Other Names: O2
  Arms: Oxygen 21%

SUMMARY:
The purpose of this study is to determine whether low concentration inhaled carbon monoxide is effective in treating idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is an interstitial lung disease characterized by destruction of normal epithelial structure, proliferation of fibroblasts, and deposition of connective-tissue matrix proteins. There are currently no effective therapies for IPF. Over the past two decades, preclinical studies of inhaled low dose carbon monoxide (CO) have shown that this biologically active diatomic gas possesses properties that would make it a viable novel therapy for IPF. CO therapy has been well tolerated in Phase I and Phase II human trials to date. This phase II study is designed to investigate whether IPF patients show evidence of decreased peripheral blood levels of matrix metalloproteinase-7 (MMP7) and stability of secondary indicators of disease progression after 3 months of inhaled therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults above the age of 18 and equal to or below the age of 85
* Diagnosis of IPF by biopsy or
* American Thoracic Society (ATS)/European Respiratory Society (ERS)/ Latin American Thoracic Association (ALAT) Guidelines (Am J Respir Crit Care Med Vol 183. pp 788-824,2011)
* Forced vital capacity (FVC) greater than or equal to 50% predicted, greater than or equal to one month off all medications prescribed for IPF

Exclusion Criteria:

* Evidence of active infection within the last month
* Significant obstructive respiratory defect
* Supplemental oxygen required to maintain an oxygen saturation over 88% at rest
* History of myocardial infarction within the last year, heart failure within the last 3 years or cardiac arrhythmia requiring drug therapy
* History of smoking within 4 weeks of screening
* Pregnancy or lactation
* Participation in another therapeutic clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-07; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosas O Ivan, MD, Principal Investigator — Brigham and Women's Hospital; Joe GN Garcia, MD, Principal Investigator — University of Illinois at Chicago
Locations (8):
- United States (8):
  - University of California San Francisco, San Francisco, California
  - University of Illinois Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University, New York, New York
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Rosas IO, Goldberg HJ, Collard HR, El-Chemaly S, Flaherty K, Hunninghake GM, Lasky JA, Lederer DJ, Machado R, Martinez FJ, Maurer R, Teller D, Noth I, Peters E, Raghu G, Garcia JGN, Choi AMK. A Phase II Clinical Trial of Low-Dose Inhaled Carbon Monoxide in Idiopathic Pulmonary Fibrosis. Chest. 2018 Jan;153(1):94-104. doi: 10.1016/j.chest.2017.09.052. Epub 2017 Oct 31. PMID 29100885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period opened on 11/29/2011 and was closed on 1/10/2014 when the study reached its enrollment target of 58 subjects. Subjects were enrolled at 8 participating academic medical centers.
Pre-assignment Details: Sixty-five subjects were screened, of which 7 subjects were screen failures. Reasons for screen failure included subjects who completed screening changed their mind about participation before visit 2, FEV1/FVC less than 70% predicted, and infection within 1 month before screening. The screening period up to 28 days from date of consent to Visit 2.
Period: Overall Study
Arm/Group | Carbon Monoxide Inhalation | Oxygen 21%
Started | 29 | 29
Completed | 22 | 23
Not Completed | 7 | 6
Not completed — Adverse Event | 6 | 2
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbon Monoxide Inhalation | Oxygen 21% | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (6.1) | 68.6 (8.4) | 68 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 25 | 22 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Serum MMP7 Level
Description: The primary study endpoint was the change in MMP7 serum concentration (ng/ml) from baseline to 12 weeks. Serum MMP7 concentrations in peripheral blood are easily measureable and reflect changes in the alveolar microenvironment. Thus, we have chosen to study mean serum MMP7 concentrations after three months of CO treatment as a surrogate biomarker of the effect of inhaled CO administration on disease progression.
Time Frame: Baseline to Week 12
Population: One subject randomized to placebo withdrew consent prior to the MMP7 blood draw at visit 2. This is missing data and the reason why we have n=28 for placebo group.
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Carbon Monoxide Inhalation | Oxygen 21%
Number analyzed (Participants) | 29 | 28
ng/ml | -0.15 (0.58) | 0.88 (0.57)
Statistical Analysis 1: Comparison: Carbon Monoxide Inhalation vs Oxygen 21%; Test type: Superiority; p = 0.2072, ANOVA; Repeated measure ANOVA; Mean Difference (Net) = -1.04, Standard Error of Mean 0.81 — Difference = (Change from baseline to Week 12 for Carbon monoxide group) minus (Change from baseline to Week 12 for Placebo group)

2. Secondary Outcome: Total Lung Capacity % Predicted Values (TLC)
Description: Total lung capacity % predicted values (TLC) is a major clinical determinant of restrictive lung disease in practice, with TLC measurement below the 5th percentile of the predicted value indicative of a restrictive ventilatory defect
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: % Predicted
Arm/Group | Carbon Monoxide Inhalation | Oxygen 21%
Number analyzed (Participants) | 29 | 29
% Predicted | -2.29 (1.12) | -1.44 (1.10)
Statistical Analysis 1: Comparison: Carbon Monoxide Inhalation vs Oxygen 21%; Test type: Superiority; p = 0.5882, ANOVA; Repeated Measure ANOVA; Mean Difference (Net) = -0.85, Standard Error of Mean 1.57 — Difference = (Change from baseline to week 12 for CO group) minus (Change from baseline to week 12 for placebo group)

3. Secondary Outcome: Diffusing Capacity for Carbon Monoxide (DLCO) % Predicted Values
Description: Interstitial changes associated with IPF can worsen diffusing capabilities across the alveolar-capillary membrane. As a result, diffusing capacity of carbon monoxide is an important outcome to assess architectural distortion and resultant decrements in diffusing capabilities
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: % predicted
Arm/Group | Carbon Monoxide Inhalation | Oxygen 21%
Number analyzed (Participants) | 29 | 29
% predicted | 1.10 (1.41) | 0.46 (1.32)
Statistical Analysis 1: Comparison: Carbon Monoxide Inhalation vs Oxygen 21%; Test type: Superiority; p = 0.7401, ANOVA; Repeated Measure ANOVA; Mean Difference (Net) = 0.64, Standard Error of Mean 1.93 — difference=(change from baseline to week 12 for CO group) minus (change from baseline to week 12 for placebo group)

4. Secondary Outcome: Six Minute Walk Distance
Description: The six minute walk distance is commonly used both in research studies and in clinical practice as a measure of functional capabilities, and changes in six minute walk distance and oxygen use during testing over time often reflect clinically relevant disease progression. We will measure the distance travelled during six minutes (meters) in accordance with published guidelines
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Carbon Monoxide Inhalation | Oxygen 21%
Number analyzed (Participants) | 29 | 29
meters | -35.54 (12.83) | 12.92 (12.83)
Statistical Analysis 1: Comparison: Carbon Monoxide Inhalation vs Oxygen 21%; Test type: Superiority or Other; p = 0.0099, ANOVA; Repeated measure ANOVA; Mean Difference (Net) = -48.46, Standard Error of Mean 18.14 — Difference=(Change from baseline to week 12 for CO group) minus (Change from baseline to week 12 for placebo group)

5. Secondary Outcome: St George's Respiratory Questionnaire
Description: St. George's Respiratory Questionnaire (SGRQ) is a validated self-reported instrument. In this instrument, scores range from 0 to 100, with higher scores reflective of worse quality of life.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Total Score
Arm/Group | Carbon Monoxide Inhalation | Oxygen 21%
Number analyzed (Participants) | 29 | 29
Total Score | -2.12 (1.70) | -1.55 (1.72)
Statistical Analysis 1: Comparison: Carbon Monoxide Inhalation vs Oxygen 21%; Test type: Superiority; p = 0.8124, ANOVA; Repeated measure ANOVA; Mean Difference (Net) = -0.58, Standard Error of Mean 2.42

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the start of treatment through 28 days after discontinuation of the study.
Arm/Group | Carbon Monoxide Inhalation | Oxygen 21%
Serious Adverse Events (participants affected / at risk) | 3/29 | 7/29
Other Adverse Events (participants affected / at risk) | 28/29 | 19/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbon Monoxide Inhalation (N=29) | Oxygen 21% (N=29)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
IPF progression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acute pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Worsening Cirrhosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute syndrome of innapropriate antidiuretic hormone (SIADH) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Small Cell Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Worsening of Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Fibrosis Related Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbon Monoxide Inhalation (N=29) | Oxygen 21% (N=29)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 2 (3)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 8 (10)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 2 (3)
Fatigue (General disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 5 (6) | 8 (9)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 4 (5) — Common Cold symptom
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No